CLINICAL TRIAL: NCT02306369
Title: Internet-delivered CBT for Irritable Bowel Syndrome in Adolescents - a Randomized Controlled Study
Brief Title: Internet-delivered CBT for Irritable Bowel Syndrome in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Brjann Ljotsson, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ibs 13-17 år 2013
Record Dates: First submitted 2014-09-08; First posted 2014-12-03 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Irritable Bowel Syndrome; Functional Gastrointestinal Disorders
Keywords: ICBT; IBS; FGID; functional abdominal pain; Adolescents; Children; Treatment; CBT; Exposure; Cognitive Behavior Therapy; Internet; Computerized; Abdominal Pain; Functional Pain; Functional Disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases; Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as usual (No Intervention): A wait-list control.
- Internetdelivered exposure-based CBT (Experimental): 10 sessions of ICBT during 10 weeks for the adolescents. 5 session of parent training during 10 weeks for parents. Therapist support is provided at least once weekly through the platform developed for the purpose. Therapists are trained CBT-psychologists.
  Interventions: Behavioral: Internetdelivered exposure-based CBT

INTERVENTIONS:
Behavioral: Internetdelivered exposure-based CBT — The Internet-delivered exposure treatment is based on the well-established internet-delivered CBT-treatment for IBS in adults, and adapted for adolescents and their parents. The feasibility of the treatment were tested in a pilot study during 2012. Components in the treatment are exposure for symptoms and parent training. The purpose of the treatment is to reduce fearful and anxious responses to symptoms and lessen avoidance of symptoms in the adolescents, and to teach the parents how parental behavior can influence symptoms in children. Detailed behaviour analysis is made for each individual and instruction is given on how to gradually expose to symptoms to lessen fear for symptoms and widen the behavioral repertoire.
  Arms: Internetdelivered exposure-based CBT

SUMMARY:
This randomized controlled trial aims to evaluate the treatment effects of an internet-delivered CBT-program for adolescents with irritable bowel syndrome.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is prevalent and associated with low quality of life in adolescents. Medical or dietary treatments lack evident efficiency, while psychosocial interventions, i.e. cognitive behavior therapy (CBT)has shown promising effects in face-to-face treatments. Therapists trained to deliver CBT for IBS are scarce, leading to a situation where very few adolescents with IBS receive the only evidence-based intervention. Exposure-based internet-delivered CBT (ICBT) for adults with IBS has shown strong stable effects and cost-efficency. Our aim is to develop a treatment that enhances the availability to evidence-based treatment for children and adolescents with IBS. Such a treatment could swiftly be implemented in regular health care for this large population. The main purpose of this study is to compare the effectiveness of exposure-based ICBT to treatment as usual (wait-list) for adolescents with IBS.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17 at inclusion date.
* fulfilling Rome III-criteria for IBS with a written statement from patient's physician confirming a diagnosis of IBS and negative required tests (Blood samples: C-reactive protein or erythrocyte sedimentation rate, Blood count and IgA-Transglutaminase. Stool: f-Calprotectin).

Exclusion Criteria:

* concurrent serious medical conditions.
* a psychiatric diagnosis, judged to be a more important treatment target than the abdominal pain.
* on-going psychological treatment.
* absence from school exceeding an average of 2 days a week is a cause for exclusion since high absence demands more intensive interventions than can be offered in ICBT.
* on-going abuse or severe parental psychiatric illness in the family.
* since treatment format assumes normal reading and writing skills, pronounced language skill deficits and learning difficulties lead to exclusion from the study.
* lack of regular internet-access.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2013-11; Primary Completion 2016-05 (Actual); Study Completion 2017-11-18 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptom Rating Scale-IBS Version (GSRS-IBS). | Baseline to 10 weeks.
  Change in gastrointestinal symptoms measured with a self-rating scale from baseline to 10 weeks for analysis of effect. The GSRS-IBS have 13 items about weekly gastrointestinal symptoms like bloating, hard stool, abdominal pain etc. It is a seven-point Likert scale from 1 (no discomfort at all) to 7 (very severe discomfort). The GSRS-IBS has excellent psychometric properties with internal consistency between α = .74 (for abdominal pain) to α = .85 (for satiety).
Gastrointestinal Symptom Rating Scale-IBS Version (GSRS-IBS). | Baseline to 9 months.
  Change in gastrointestinal symptoms measured with a self-rating scale from baseline to 9 months for analysis of effect. The GSRS-IBS have 13 items about weekly gastrointestinal symptoms like bloating, hard stool, abdominal pain etc. It is a seven-point Likert scale from 1 (no discomfort at all) to 7 (very severe discomfort). The GSRS-IBS has excellent psychometric properties with internal consistency between α = .74 (for abdominal pain) to α = .85 (for satiety).
Gastrointestinal Symptom Rating Scale-IBS Version (GSRS-IBS). | Baseline to 15 months.
  Change in gastrointestinal symptoms measured with a self-rating scale from baseline to 15 months baseline for analysis of effect. The GSRS-IBS have 13 items about weekly gastrointestinal symptoms like bloating, hard stool, abdominal pain etc. It is a seven-point Likert scale from 1 (no discomfort at all) to 7 (very severe discomfort). The GSRS-IBS has excellent psychometric properties with internal consistency between α = .74 (for abdominal pain) to α = .85 (for satiety).
Gastrointestinal Symptom Rating Scale-IBS Version (GSRS-IBS). | Baseline to 27 months.
  Change in gastrointestinal symptoms measured with a self-rating scale from baseline to 27 months for analysis of effect. The GSRS-IBS have 13 items about weekly gastrointestinal symptoms like bloating, hard stool, abdominal pain etc. It is a seven-point Likert scale from 1 (no discomfort at all) to 7 (very severe discomfort). The GSRS-IBS has excellent psychometric properties with internal consistency between α = .74 (for abdominal pain) to α = .85 (for satiety).

SECONDARY OUTCOMES:
Faces pain scale - R | Weekly during treatment (treatment week 1-9). Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in pain intensity measured with a self-rating scale weekly during treatment for mediation analyses, and from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months for analysis of effect.The Faces Pain Scale is a self-report measure used to assess the intensity of children's pain. Faces have four faces representing least pain and most pain on equal intervals on a scale from 0-10. Its validity is supported by a strong positive correlation (r=0.93, N=76) with a visual analogue scale (VAS) measure in children aged 5-12 years. The metric for scoring (0-10) conforms closely to a linear interval scale.
IBS-behavioral responses questionnaire (IBS-BRQ). | Weekly during treatment (treatment week 1-9). Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in IBS-specific behaviors measured with a self-rating scale weekly during treatment for mediation analyses, and from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months for analysis of effect. IBS-BRQ is a self-rating scale measuring IBS-specific behavioral responses shown to be unhelpful and probably maintain IBS-symptoms. The scale consists of 26 items on a seven-point Likert scale from 1 (never) to 7 (always). The scale includes items related to avoidance behavior such as "I avoid certain social situations (e.g. restaurants) because of my IBS" and to toilet behavior such as "I spend more time on the toilet than ideally I would like". IBS-BRQ is both reliable and valid with a high degree of internal consistency for adults with IBS (Cronbach's α=.86). The scale differentiate significantly between IBS patients and healthy controls (F=221, P<.01).
Percieved Stress scale (PSS 10) | Weekly during treatment (treatment week 1-9). Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in perceived stress measured with a self-rating scale weekly during treatment for mediation analyses, and from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months for analysis of effect. The PSS measures the degree to which situations are appraised as stressful. It is a self-report scale with 10 items on daily hassles and the current feeling of being able to handle problems that need to be addressed. It is a five-point Likert scale ranging from 0 (never) to 4 (very often). It is a widely used questionnaire to measure perceived stress and has adequate internal and test-retest reliability.
Pain reactivity Scale (PRS) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in pain reactivity measured with a self-report scale, pain reactivity scale (PRS), at baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months. PRS have 5 items about reactivity to and worry about pain. Three items are about emotional reactions to current pain. Two items affect frequency of worry about not being able to do things now, and in the future because of the pain. Questions are answered on a 6-point scale from 0 ("not at all") to 6 ("very much"). PRS has been reported to have satisfactory psychometric properties (Wicksell et al, 2011)
Pain interference index (PII) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in pain interference measured with a self-report scale at baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months. Pain interference index (PII), have 6 items about interference on various activities because of pain. Questions are answered on a 6-point scale from 0 ("not at all") to 6 ("very much"). According to preliminary analysis, the instrument has satisfactory psychometric properties (Wicksell et al., 2011)
Functional disability index (FDI) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in function measured with a self-report scale at baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months. Functional disability index (FDI) have15 items on daily activities. Questions are related to specific activities such as climbing stairs, running 100 meters and to go shopping, and general activities such as eating meals and being in school all day. The scale ranges from 1 (no problem at all) to 5 (impossible). It is validated for children and adolescents with chronic abdominal pain with high internal consistency, α = .86 for boys and α = .91 for girls (Claar and Walker, 2006). FDI is the scale that is recommended in pediatric pain studies to measure the influence of pain on function (McGrath et al., 2008).
Visceral sensitivity Index (IBS-VSI) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in visceral sensitivity from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months measured with a self-report scale that measures gastrointestinal symptom-specific anxiety. VSI is a 15-item scale and has a scale ranging from 0 (not at all) to 5 (totally agree). The scale has demonstrated excellent reliability as well as good content, convergent, divergent and predictive validity.
Gastrointestinal Symptom Rating Scale-IBS Version (GSRS-IBS). | Weekly during treatment (treatment week 1-9).
  Change in gastrointestinal symptoms measured weekly with a self-rating scale during treatment for mediation analyses. The GSRS-IBS have 13 items about weekly gastrointestinal symptoms like bloating, hard stool, abdominal pain etc. It is a seven-point Likert scale from 1 (no discomfort at all) to 7 (very severe discomfort). The GSRS-IBS has excellent psychometric properties with internal consistency between α = .74 (for abdominal pain) to α = .85 (for satiety).
Pediatric Quality of Life Inventory (PedsQL) Generic Core scales age 13-18 | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in quality of life from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months measured with a self-report scale that measures quality of life in adolescents. PedsQL Generic Core scales is a 23-item scale ranging from 0 (never) to 4 (almost always). The PedsQL is shown to distinguishe between healthy children and adolescents and pediatric patients with acute or chronic health conditions and demonstrate acceptable reliability and validity.
Pediatric Quality of Life Inventory (PedsQL) Gastrointestinal Symptom Scale | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in gastrointestinal symptoms from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months measured with a self-report scale that measures gastrointestinal symptoms in children and adolescents. The PedsQL Gastro is a 9-item scale ranging from 0 (never) to 4 (almost always).
Children´s Somatization Inventory (CSI-24) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in inner symptoms from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months measured with a self-report scale that measures inner symptoms (e.g., headache, nausea, heart racing) that often, but not necessarily, occur in the absence of identified disease, in children and adolescents. CSI-24 is a 24-item scale ranging from ranging from 0 '(not at all) to 4 (a whole lot).
Spence Children's Anxiety Scale (SCAS-C) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in anxiety symptoms from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months measured with a self-report scale that measures anxiety symptoms in children and adolescents. SCAS-C is a 45 -item scale ranging from ranging from 0 (never) to 3 (always). SCAS-C has demonstrated high internal consistency, high concurrent validity with other measures of child and adolescent anxiety, and adequate test-retest reliability.
TiC-P Adolescents revised version | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in healthcare utilization and productivity loss from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months measured with a self-report scale that measures healthcare utilization and productivity. The scale has been revised to fit adolescents and consists in our study of 3 items assessing school absenteeism and 6 items assessing healthcare utilization.
TIC-P Parent report | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in parents healthcare utilization and productivity loss from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months measured with a self-report scale that measures healthcare utilization and productivity. TIC-P consists of 10 items.
Generalized Anxiety Disorder Screener (GAD-7) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in anxiety levels in parents from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months measured with a self-report scale that measures anxiety symptoms. GAD-7 is a 7-item scale ranging from 0 (not at all) to 3 (almost every day). Evidence supports reliability and validity of the GAD-7 as a measure of anxiety in the general population.
Patient Health Questionnaire (PHQ 9) | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in depression levels in parents from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months measured with a self-report scale that measures depression. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). PHQ-9 is shown to be a reliable and valid measure of depression severity in adults.
ARCS | Baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months.
  Change in parents responses to their children's abdominal pain from baseline to 10 weeks, baseline to 9 months, baseline to 15 months, baseline to 27 months measured with a self-report scale assessing protectiveness, minimizing, and encouraging responses to children's pain behavior. The ARCS is a 29-item scale.

CONTACTS AND LOCATIONS:
Overall Officials: Brjánn Ljótsson, PhD, Principal Investigator — Departement of Clinical neuropsychology, Karolinska Institutet
Locations (1):
- Child and Adolescent Psychiatry (CAP) Research Center, Stockholm, County of Stockholm, Sweden

REFERENCES:
- [Derived] Sampaio F, Bonnert M, Olen O, Hedman E, Lalouni M, Lenhard F, Ljotsson B, Ssegonja R, Serlachius E, Feldman I. Cost-effectiveness of internet-delivered cognitive-behavioural therapy for adolescents with irritable bowel syndrome. BMJ Open. 2019 Jan 24;9(1):e023881. doi: 10.1136/bmjopen-2018-023881. PMID 30679293